CLINICAL TRIAL: NCT00753168
Title: A Randomized, Parallel-Group, Multi-Center, Investigator-Masked, Active-and Placebo-Controlled, Phase 1-2 Evaluation of the Safety and Efficacy of OT-730 Ophthalmic Solution in Reducing the Intraocular Pressure in Subjects With Ocular Hypertension or Open-Angle Glaucoma
Brief Title: Phase 1-2 Evaluation of OT-730 Eye Drops in Reducing the Intraocular Pressure in Patients With Ocular Hypertension or Open-Angle Glaucoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Othera Pharmaceuticals (Industry)
Responsible Party: Alison Brown, Othera Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OT-730-C01
Record Dates: First submitted 2008-09-08; First posted 2008-09-16 (Estimated); Last update posted 2009-01-07 (Estimated); Status verified 2009-01

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
Keywords: glaucoma, open angle, ocular hypertension, beta blocker, beta adrenergic, intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): OT-730 ophthalmic solution
  Interventions: Drug: OT-730 ophthalmic solution
- 2 (Active Comparator): timolol maleate ophthalmic solution
  Interventions: Drug: timolol maleate ophthalmic solution
- 3 (Placebo Comparator): placebo eye drops
  Interventions: Drug: OT-730 placebo

INTERVENTIONS:
Drug: OT-730 ophthalmic solution — one eye drop twice daily
  Arms: 1
Drug: timolol maleate ophthalmic solution — one eye drop twice daily
  Arms: 2
Drug: OT-730 placebo — one eye drop twice daily
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the safety and potential efficacy of a new drug, OT-730 ophthalmic solution (eye drops), in reducing intraocular pressure in the eyes of patients with open angle glaucoma or ocular hypertension. It will be compared with commercial timolol and placebo eye drops.

DETAILED DESCRIPTION:
Glaucoma is a group of diseases of the eye that can result in irreversible vision loss due to damage to the optic nerve. Elevated intraocular pressure (IOP) is one factor associated with glaucoma. Currently-available medication used to lower IOP includes beta-blocking agents, which can have undesirable side effects on the cardiac and respiratory systems.

The OT-730 ophthalmic solution contains OT-730, a prodrug that, when applied as an eyedrop, metabolizes to OT-705, an active beta blocker. The OT-730 ophthalmic solution is being studied to see how well it lowers IOP in patients with a diagnosis of open angle glaucoma or ocular hypertension. It will be compared with a well known beta blocker, timolol maleate ophthalmic solution, and with a placebo eye drop, in order to assess its ability to lower IOP without the typical side effects of other beta blockers.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects, 18 to 80 years of age, any gender
* diagnosis of primary open angle, pseudoexfoliative or pigmentary glaucoma or ocular hypertension

Exclusion Criteria:

* have VA worse than 20/200,
* cataract that compromises visualization of fundus,
* history of lack of response to ocular beta blocker therapy,
* uncontrolled intraocular pressure,
* angle closure glaucoma or occludable angles,
* retinal detachment, macular hole, progressive vision loss, any progressive retinal disease or neurologic disease other than glaucoma that is likely to worsen visual field or acuity during the course of the study,
* a history of, or any current condition contraindicated with use of a beta blocker (e.g., chronic obstructive pulmonary disease, bronchial asthma, congestive heart failure, myasthenia gravis, hypoglycemia, bradycardia, etc),
* chronic use of steroids,
* any disease that, in the opinion of the investigator, may put the patient at significant risk,
* taking systemic beta blockers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Assess the safety profile of OT-730 | 8 days
Change from baseline in intraocular pressure | Day 6

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Artesia, California
  - Roswell, Georgia
  - Charlotte, North Carolina
  - High Point, North Carolina
  - Mt. Pleasant, South Carolina

REFERENCES:
- See also: Othera Pharmaceuticals, Inc. website — http://www.othera.com